CLINICAL TRIAL: NCT03184883
Title: Comparative Study of Conventional Versus Flexible Mandibular Single Complete Denture
Brief Title: Comparative Study Between Acrylic and Flexible Dentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marianne Azer, Comparative Study of Conventional versus Flexible Mandibular Single Complete Denture, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: evidence committee
Record Dates: First submitted 2017-06-02; First posted 2017-06-14 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single conventional denture (Experimental): patients with mandibular edentulous arch by using acrylic resin denture with soft linner
  Interventions: Procedure: single conventional denture
- single flexible denture (Active Comparator): patients with mandibular edentulous arch by using flexible lower denture
  Interventions: Procedure: single flexible denture

INTERVENTIONS:
Procedure: single conventional denture — mandibular conventional denture with soft liner
  Arms: single conventional denture
Procedure: single flexible denture — mandibular flexible compete denture
  Arms: single flexible denture

SUMMARY:
comparing the effect of conventional mandibular single denture with flexible mandibular single denture on tissue and patient's satisfaction

DETAILED DESCRIPTION:
comparing the effect of conventional mandibular single denture with flexible mandibular single denture on tissue by keratinization index through PAP stain and patient's satisfaction through a questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Mandibular flat ridge
2. Patient with opposing natural teeth or satisfactory fixed prostheses
3. Angle class I Maxillimandibular relationship
4. No intraoral soft and hard tissue pathosis
5. Non smokers
6. Patients with no previous denture experience
7. Patients having last extraction at least 6 month before denture construction

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Cytological changes manifested as keratinization index | 6 months
  Objective Outcome: measuring the cytological changes manifested as keratinization index

CONTACTS AND LOCATIONS:
Overall Officials: Essam Aziz, professor, Principal Investigator — supervisor

IPD SHARING:
Plan to Share IPD: No